CLINICAL TRIAL: NCT04558385
Title: Seroconversion in COVID-19 Recovered Population: an Observational Study
Brief Title: Seroconversion in COVID-19 Recovered Population
Status: Completed | Type: Observational
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Amina Asif, Assistant Professor, Lahore General Hospital
Other Study IDs: LGH006
Record Dates: First submitted 2020-09-20; First posted 2020-09-22 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IgG SARS CoV2 — IgG SARS CoV 2 will be checked in serum of COVID 19 recovered population

SUMMARY:
This study investigate the kinetics of IgG responses to both N and S proteins in the subjects who suffered from COVID 19 and then had recovered.

DETAILED DESCRIPTION:
Coronaviruses (CoVs) are enveloped, single positive-strand RNA viruses belonging to the large subfamily Coronavirinae, which can infect mammals and several other animals.The continued spread of coronavirus disease 2019 (COVID-19) has prompted widespread concern around the world, and the World Health Organization (WHO), on 11 March 2020, declared COVID-19 a pandemic. Studies on severe acute respiratory syndrome (SARS) and Middle East respiratory syndrome (MERS) showed that virus-specific antibodies were detectable in 80-100% of patients at 2 weeks after symptom onset. Currently, the antibody responses against SARS-CoV-2 remain poorly understood and the clinical utility of serological testing is unclear Little is known about the kinetics, tissue distribution, cross-reactivity and neutralization antibody response in COVID-19 patients .

The seropositivity rate of both IgM and IgG responses after onset and recovery of disease, and in the context of both N protein and S protein has not been clarified. The kinetics of antibody responses in critical cases or ICU patients has not been reported, and no studies have suggested whether antibody response is associated with disease prognosis

ELIGIBILITY:
Inclusion Criteria:

Subjects recovered from COVID 19 confirmed on PCR or clinically

Exclusion Criteria:

subjects who have not been confirmed suffering from COVID 19 by PCR or clinically

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: population who have suffered from COVID 19, whose disease was either confirmed by PCR or clinically and then recovered
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
IgG SARS CoV2 | 5 months
  Presence or absence of SARV CoV2 IgG antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Amina Asif, MPhilMicro, Principal Investigator — LahoreGeneralHospital.Lahore
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided